CLINICAL TRIAL: NCT05171868
Title: Eye Movement Desensitization and Reprocessing (EMDR) for Stress, Psychological Trauma and Suicidal Ideation in Police Personnel: A Feasibility Randomised Controlled Trial
Brief Title: Eye Movement Desensitization and Reprocessing (EMDR) for Police Personnel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHAR M-EMDR-001
Record Dates: First submitted 2021-12-11; First posted 2021-12-29 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Suicidal Ideation; Psychological Trauma; Stress
Keywords: Forensic settings; EMDR; Trauma; Police Personnel; Suicidal Ideation; Stress; Pakistan; Feasibility
MeSH Terms: conditions — Suicidal Ideation; Psychological Trauma; Wounds and Injuries | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR receiving group (Experimental): EMDR is a psychotherapeutic approach that emphasizes the role of the brain's information processing system in perfecting the psychological consequences of distressing events. EMDR is an eight-phase treatment protocol, including procedure that focuses on the memories underlying current problems and those that must be specifically addressed to bring the client to a robust state of psychological health. One of its distinguishing aspects is its use of bilateral physical stimulation, such as side-to-side eye movements, alternating hand taps, or alternating auditory tones while the person undergoing treatment is mentally focusing on aspects of various life experiences.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing (EMDR)
- Waiting list Control Group (No Intervention): The control group will receive their routine care as usual. Once the trial is completed they will be invited for EMDR sessions

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) — Each participant in the intervention group will receive 8 individual, weekly EMDR sessions over 8 weeks. Each session will take approximately 60-90 minutes. The sessions will be delivered at a place convenient to the participant. Trained EMDR therapists will deliver the intervention.
  Arms: EMDR receiving group

SUMMARY:
Objectives:

1. To examine the feasibility of Eye Movement Desensitization and Reprocessing (EMDR) as an intervention to reduce psychological trauma and stress amongst police officers in Pakistan.
2. To test whether reducing stress and psychological trauma reduces suicidal ideation in police officers.
3. To explore participants' experiences with EMDR Intervention.

Study design and setting:

The study will be a mixed-method feasibility randomized controlled trial of EMDR as an intervention in treating symptoms such as stress, trauma and suicidal ideation in police officers. The study will be conducted in five major cities in Pakistan: Rawalpindi, Karachi, Peshawar, Quetta, and Lahore.

Sample size:

A total of N=80 eligible police officers will be recruited and randomized in the study.

DETAILED DESCRIPTION:
EMDR intervention is an evidence-based psychological intervention that has been proven effective for stress and trauma, however, research evidence on feasibility of EMDR in forensic settings in Pakistan is limited. The current study aims to establish the feasibility and acceptability of EMDR intervention for management of stress, psychological trauma and suicidal ideation amongst police officers in Pakistan. The study will recruit a total of 80 police officers from police stations in the participating study sites, and prospective participants will be screened against eligibility criteria. Eligible consented participants will be enrolled in the study. An independent statistician will randomize participants to one of the two study arms: 1) EMDR (Intervention); or 2) waiting list control arm. Each participant in the intervention arm will receive 8 individual, weekly EMDR sessions over 8 weeks. Each session will take approximately 60-90 minutes. The sessions will be delivered at a place convenient to the participants. Trained EMDR therapists will deliver the intervention. The waiting list control arm will receive their routine care as usual, As part of the safety protocol, the details of any services each participant receives in the control group will be obtained. EMDR treatment will be offered to the control group (waiting control group) after the active intervention is complete. Assessment measures will be administered before and after the intervention at 8th week. All assessments will be rater blind. After post-assessments at 8th week, a purposefully selected subset (stratified by age & gender) of participants will be invited for qualitative interviews to explore their experiences and satisfaction with the intervention. Participants will be interviewed within 1 week of their post-intervention by a trained qualitative researcher exploring their experience with EMDR, the barriers and facilitators to engagement, and perceived benefits or negative experiences with the intervention. A sample of up to 15 interviews would be enough to achieve category saturation. On average, interviews will last for 60 minutes. The interview will be face-to-face or through telephone as an alternative to a face-to-face meeting to reduce the number of in-person meetings given the current context of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Having suicidal ideation measured as a score > 2 on Beck scale of suicidal ideation
* Aged 18 years - 60 years' old
* Police officer with psychological trauma measured with the International Trauma Questionnaire and stress measured with stress subscale of Depression, Anxiety and Stress scale

Exclusion Criteria:

* Less than 12 months' experience in the police officer.
* Participants reporting active suicidal ideation measured as a score of 2 on item no 4 of BSSI will be excluded and referred to a psychiatric service.
* With current history of use of hard/psychoactive substances (excluding tobacco and caffeine).
* Unable to provide consent due to severe mental or physical illness.
* Unlikely to be available for the entire duration of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | From baseline to 8th week (at the end of intervention)
  The feasibility will be determined by collecting data on recruitment rates. The success criterion of feasibility will be to recruit > 50% of eligible participants.
Acceptability measure | From baseline to 8th week (at the end of intervention)
  Intervention acceptability will be assessed using data on intervention attendance. The criterion for acceptability is the intervention attendance rate of > 5 sessions.
Feasibility of Retention | From baseline to 8th week (at the end of intervention)
  The feasibility of retention will be determined by collecting data on retention rates. The success criterion of feasibility of retention will be to retain > 50% participants.

SECONDARY OUTCOMES:
Beck Scale for Suicide Ideation | Change in problem scores from baseline to 8th week
  Beck Scale for Suicide Ideation is a 19-item instrument for detecting and measuring the current intensity of patient-specific attitude, behavior, and specificity of patient thoughts to kill themselves during the past week.
The International Trauma Questionnaire | Change in problem scores from baseline to 8th week
  The International Trauma Questionnaire is a brief, simple-worded measure focusing on the core features of post-traumatic stress disorder.
Depression Anxiety and Stress Scale | Change in problem scores from baseline to 8th week
  Depression Anxiety and Stress Scale is consist of three subscales that measure the negative emotional states of depression, anxiety, and stress and consist of 7 items per subscale. The participants are requested to use 4-point severity/frequency scales to rate the extent to which they have experienced each state over the past week.
Beck Hopelessness Scale | Change in problem scores from baseline to 8th week
  Beck hopelessness scale measure three aspects of hopelessness; feelings about the future, loss of motivation and expectations. The scale consists of 20 statements each of which is scored as 0 or 1.
Sleep Quality Questionnaire | Change in problem scores from baseline to 8th week
  Sleep Quality Questionnaire consists of eight items rated on a 5-point scale. It measures self-reported alertness, sleepiness, tiredness, and functional impairments associated with sleep and problems during waking hours within the past seven days.
Coping Resource Inventory | Change in coping resources scores from baseline to 8th week
  The Coping Resource Inventory assesses the individual's stress management and coping resources with stress.

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husain, Principal Investigator — University of Manchester; Nasim Chahudhry, Principal Investigator — Pakistan Institute of Living and Learning
Locations (1):
- Prison settings Peshawar, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No